CLINICAL TRIAL: NCT04587440
Title: Is the Dynamic of the Pelvic Bone Altered After a Total Hip Replacement ?
Acronym: DYPAMAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 29BRC20.0120
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Coxarthrosis; Primary; Coxarthrosis; Secondary
MeSH Terms: conditions — Osteoarthritis, Hip; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Study of the variation of the dynamic of the pelvic bone in pre and post operative of a hip replacement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient (Experimental): All patients will have a clinical examination before surgery and another 3 months after surgery, each including :
  * A medical examination
  * 3 pelvic inclination measurements (1 sitting, 1 lying and 1 standing). These measurements will be done by ultrasound devices.
  * 2 EOS X-rays (1 standing and 1 sitting) of the lower limbs and spine
  * Harris hip score
  * Pain quantification thanks to an EVA scale
  * hand-ground distance
  Interventions: Other: Pelvic inclination measurement

INTERVENTIONS:
Other: Pelvic inclination measurement — Ultra-sound based measurements of the pelvic inclination lying, standing and seating position. EOX X-ray in seating position.

SUMMARY:
Total hip replacement is one of the most common surgical procedure in France. In 2010, an estimated 147 513 total hip procedures were performed. This number is constantly increasing.

Although it is common, it can lead to many complications. The intra-prosthetic luxation is the second one after aseptic loosening.

The luxation risk is multifactorial and depends on the relative orientation of femoral et acetabular components. This orientation is influenced by statics and dynamics parameters.

So far, the literature shows that only static parameters are considered by surgeons. Thus, in reference to Lewinneck publication, which states that the luxation risk is lower if the cup is oriented with 15° +/- 10° of anteversion and 40°+/- 10° of inclination with respect to the anterior pelvic plan (APP). Defined by the two anterosuperior iliacs spines and pubic symphysis.

However, this approach is only static and do not take into account the variations of pelvic plan orientation during everyday life.

To consider these variations of pelvic inclination, it is possible to measure the angle between APP and the horizontal (in lying position) or the vertical (in standing position) plan.

Several devices allow the measure of pelvic inclination but they all have important limits (EOS radiography, scanner or navigation). A new device has been developed in Brest to measure this inclination in several positions of the daily life.This software has already been tested in healthy volunteers and results demonstrate an excellent accuracy and reproducibility.

The goal of this study is to described the dynamic of the pelvic bone thanks to this ultrasound based device, and to assess the amount of variation induced by hip replacement procedures.

ELIGIBILITY:
Inclusion criteria :

* Patient with primary or secondary hip arthritis, at stage II to III of the radiological classification of Tönnis and for whom total hip replacement is indicated by surgeon.
* Signed consent
* Patient beneficiary of a social security plan

Exclusion Criteria:

* Patient Under 18
* Patient Under protective measure (guardianship, curatorship) or unable to consent
* Patient requiring revision THR
* Patient with geographic mobility plan before the end of the follow-up
* Symptomatic contralateral hip
* Symptomatic dorsolumbar rachis
* Pelvis or spine surgery planed during the follow-up
* Pregnant or nursing woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2023-02-02 (Estimated); Study Completion 2023-08-02 (Estimated)

PRIMARY OUTCOMES:
Variation of the pelvic incidence | Day 0 - Month 3
  The main evaluation criterion is the variation of the pelvic incidence between pre- and post-operative total hip replacements

SECONDARY OUTCOMES:
Analysis of the correlation between the variation in pelvic incidence while sitting, standing and lying down and the implant settings | Day 0 - Month 3
  Assessed by EOS X-Ray.
Analysis of the correlation between variation in pelvic incidence while sitting, standing and lying down and clinical parameters (Harris hip score) | Day 0 - Month 3
  Clinical examination (Harris hip score) will be performed at day 0 and month 3.
Analysis of the correlation between variation in pelvic incidence while sitting, standing and lying down and clinical parameters (EVA) | Day 0 - Month 3
  Clinical examination (EVA) will be performed at day 0 and month 3.
Analysis of the correlation between variation in pelvic incidence while sitting, standing and lying down and clinical parameters (Hand-ground distance) | Day 0 - Month 3
  Clinical examination (Hand-ground distance) will be performed at day 0 and month 3.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion.
Access Criteria: Data access request will be reviewed by the internal committee of Brest University Hospital. Requestor will be required to sign and complete a data access agreement.